CLINICAL TRIAL: NCT01580618
Title: TNK for Loculated Pleural Effusions in Patients With Malignancy
Brief Title: Tenecteplase (TNK) for Loculated Pleural Effusions in Patients With Malignancy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unable to accrue patients at a reasonable rate
Sponsor: Kaiser Permanente (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Hyo-Chun Yoon, Staff Radiologist, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HI-07HYoon-02
Record Dates: First submitted 2010-09-17; First posted 2012-04-19 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Pleural Effusion
Keywords: pleural effusion; malignancy; loculated
MeSH Terms: conditions — Pleural Effusion; Neoplasms | interventions — Saline Solution; Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Placebo Comparator): Loculated pleural effusion infused with normal saline twice a day for three days.
  Interventions: Drug: normal saline
- TNKase (Active Comparator): Loculated pleural effusion infused with TNK twice a day for three days.
  Interventions: Drug: TNK (Tenecteplase)

INTERVENTIONS:
Drug: normal saline — Injection of 60 ml normal saline twice a day for three days using the existing chest tube.
  Arms: Normal Saline
Drug: TNK (Tenecteplase) — Injection of 4 mg of TNK with 59 ml normal saline into the existing chest tube twice a day for three days.
  Other Names: TNKase, tenecteplase
  Arms: TNKase

SUMMARY:
The objective of the study is to determine the safety and efficacy of TNK infusion for the treatment of loculated pleural effusions in patients with known malignancy compared to normal saline infusion.

DETAILED DESCRIPTION:
The design of the trial will be as a single-center, prospective, blinded, randomized trial comparing the infusion of TNKase versus saline for treatment of symptomatic loculated pleural effusion in patients with malignancy. Patients with known malignancy and symptomatic loculated pleural effusion who are referred for percutaneous drainage will be eligible for this study. Patients will undergo standard placement of a 8-10 french percutaneous drain into their pleural space under computed tomography or ultrasound guidance. If there is incomplete drainage of the pleural fluid at the time of initial catheter placement or if followup chest radiography performed within 24-48 hours of chest tube placement reveals persistent pleural fluid, the effusion will be considered to be loculated. After informed consent, patients will be alternately randomized to a 3 day course of twice a day intrapleural TNKase or sterile saline injections. Both the patient and the patient's primary care physician will be blinded as to the infusate. The test fluid will be kept with the pleural space for a minimum of 2 hrs before the drainage tube is returned to suction. The standard dose of TNKase will be 4 mg/60 ml NS. The control group will received 60 ml NS for each infusion. There will be a cross-over design so that patients who fail to have significant drainage during the first 2 days of therapy may be switched to the other infusate for up to an additional three days (at the primary care provider's discretion). Thus, patients who are in the saline arm will be switched to TNKase if there is a symptomatic persistent residual loculated effusion and those who fail TNKase will be switched to saline after 2 days. This is necessary in order for primary care providers to allow their patients to be enrolled in this study since our standard of care is to use Activase. We will use a cutoff of 2 days rather than 3 days before switching therapy because we cannot justify the expense of keeping patients hospitalized for an extra day in the face of failed therapy given the extremely high cost of hospitalization. Therefore, if patients have not had significant drainage in the first 2 days of therapy with either agent (saline or TNKase), the primary care provider may request that the patient be crossed over to the other agent. However, if there is some, albeit incomplete, drainage in the first 2 days of therapy, we will ask the primary care provider to wait until a complete course of intrapleural injections has been performed. We expect to enroll 40 patients during a period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age > 18 years
* Adult, non-gravid patients with malignancy and symptomatic loculated pleural effusion who has undergone percutaneous drainage will be eligible to participate. A loculated effusion is defined as an effusion whose contents cannot be completely drained at the time of initial catheter placement as documented by the initial imaging guided procedure or within 48 hours of catheter placement by chest radiography. Malignant cells need not be found within the pleural fluid.

Exclusion Criteria:

* Active internal bleeding, involving intracranial and retroperitoneal sites, or the gastrointestinal, genitourinary, or respiratory tracts
* History of stroke within 3 months
* Intracranial neoplasm, arteriovenous malformation, or aneurysm.
* Uncorrectable bleeding diathesis (INR > 1.5 despite therapy)
* Recent intracranial or intraspinal surgery or trauma
* Pregnancy (positive pregnancy test)
* Severe uncontrolled hypertension
* Documented empyema
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Participation in another clinical investigation within previous 30 days of catheter placement
* Prior enrollment in the study
* Known allergy to TNK or any of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Chun Yoon, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Foundation Hospital, Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were hospitalized patients with symptomatic loculated effusions. Each patient had a chest tube placed and loculated nature of the effusion confirmed by chest xray or CT after initial drainage of fluid from the chest tube.
Pre-assignment Details: Once loculation was documented, each patient was randomized to receive either normal saline or TNKase administered through the chest tube on a twice a day regimen for 3 days. For those in the TNKase group, each patient received 4mg TNKase in 60 mL normal saline twice daily. The normal saline group, each patient received 60mL normal saline.
Period: Overall Study
Arm/Group | Normal Saline | TNKase
Started | 8 | 12
Completed | 7 (One patient was switched from the normal saline to TNKase arm at attending physician request.) | 12
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | TNKase | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 10
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (11) | 62 (12) | 66 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Complete or Near Complete Drainage of Loculated Pleural Effusion as Determined From Chest Radiography After Three Days or Five Days of Intrapleural Therapy.
Time Frame: 3-5 days
Measure: Number; unit: percentage of participants
Arm/Group | Normal Saline | TNKase
Number analyzed (Participants) | 8 | 12
percentage of participants | 12.5 | 75

2. Primary Outcome: Percentage of Patients With Hemorrhagic Complications Associated With Catheter Drainage
Description: This is the percentage of patients in each arm of the study (Normal saline or TNKase) who suffered a hemorrhagic complication directly associated with instillation of normal saline or TNKase
Time Frame: 3-5 days
Measure: Number; unit: percentage of participants
Arm/Group | Normal Saline | TNKase
Number analyzed (Participants) | 8 | 12
percentage of participants | 12.5 | 0

3. Secondary Outcome: Percentage of Patients Who Fail Initial Therapy (TNK or Saline) Who at the Request of the Hospital-based Doctor Are Then Switched to the Other Arm/Group AND Who Then Achieve Satisfactory Drainage (Saline or TNK) Therapy.
Description: Only one patient who was on normal saline arm/group was switched (by request of the referring hospital-based doctor) to TNKase, but did not have complete clearing of their effusion. No patient in the TNKase arm/group was switched to normal saline. Therefore, we have removed the TNKase arm/group from this portion of the analysis since there are no participants in this group to analyze this outcome measure.
Time Frame: 3-5 days
Measure: Number; unit: percentage of participants
Arm/Group | Normal Saline
Number analyzed (Participants) | 1
percentage of participants | 0

4. Secondary Outcome: Percentage of Patients Able to Undergo Pleurodesis to Prevent Recurrent Pleural Effusion.
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | Normal Saline | TNKase
Number analyzed (Participants) | 8 | 12
percentage of participants | 25 | 92

5. Secondary Outcome: Duration of Hospital Stay From the Time of Initiation of Infusion Therapy for the Loculated Effusion
Description: This measures the number of hospital days for each participant after they were started on their infusion therapy.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Normal Saline | TNKase
Number analyzed (Participants) | 8 | 12
days | 13.4 (6.8) | 10.9 (4.5)

ADVERSE EVENTS:
Time Frame: From time of randomization until the time of pleural catheter removal.
Description: Intrapleural hemorrhage was the specific adverse event which can be directly related to the presence of a chest tube and/or infusion of fluid into the pleural space.
Arm/Group | Normal Saline | TNKase
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/13
Other Adverse Events (participants affected / at risk) | 0/7 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Saline (N=7) | TNKase (N=13)
intrapleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — bleeding into the pleural space from infusion of normal saline or TNKase through the existing pleural catheter

LIMITATIONS AND CAVEATS:
Results are limited due to the small numbers of patients enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes